CLINICAL TRIAL: NCT03793725
Title: A Phase II , Open-label , Investigator-initiated Trail of An Anti-PD-1 Inhibitor SHR-1210 in Combination With Apatinib in Patients With Unresectable Hepatocellular Carcinoma
Brief Title: A Trial of SHR-1210 in Combination With Apatinib in Patients With Unresectable HCC
Acronym: HZ-T-PD1-APA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yanqiao Zhang (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Yanqiao Zhang, Director of the hospital, Harbin Medical University
Organization: Harbin Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HZ-T-PD1-APA
Record Dates: First submitted 2019-01-03; First posted 2019-01-04 (Actual); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — camrelizumab; apatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-1210 + Apatinib (Experimental): Drug: SHR-1210 SHR-1210 was administered 200mg iv every 2 weeks Drug: Apatinib Apatinib was administered 500mg oral daily during the first 2 weeks and then 250 mg qd
  Interventions: Drug: SHR1210; Drug: Apatinib

INTERVENTIONS:
Drug: SHR1210 — Anti-PD-1 Antibody
Drug: Apatinib — Anti-angiogenic drugs

SUMMARY:
This is a Phase II , Open-label , Investigator-initiated Trail of SHR-1210 (an Anti-PD-1 Inhibitor) in Combination With Apatinib in Patients With unresectable Hepatocellular Carcinoma.

This study aims to evaluate the safety and efficacy of SHR-1210 combination with Apatinib as a preoperative treatment of unresectable HCC.

ELIGIBILITY:
Inclusion Criteria:

* Subjects voluntarily participate in this study and sign informed consent .
* Men or women aged 18-75 years
* patients with Unresectable HCC confirmed histologically or cytologically or clinically，At least one measurable lesion that meets the RECIST v1.1 criteria without local treatment.
* The patients can swallow pills normally.
* ECOG score was 0 or 1.
* Have a life expectancy of at least 12 weeks.
* The functions of vital organs meet the following requirements (excluding the use of any blood components and cytokines during screening) : Neutrophils≥1.5 x 109/L, Hb≥9g/dL; Plt≥90 x 109/L, ALB≥3g/dL, TSH≤ULN(Upper Limit Of Norma), TBIL ≤ 1.25 x ULN, ALT and AST ≤ 1.5 x ULN, AKP≤ 2.5 x ULN, CR≤ 1.5 x ULN
* Female Subjects of childbearing potential must have a negative serum pregnancy test within 72 hours before the first dose and must be willing to use very efficient barrier methods of contraception for the course of the study through 3 months after the last dose of study treatment.

Exclusion Criteria:

* Subjects had any active autoimmune disease or history of autoimmune disease.
* Subjects are using immunosuppressive agents, or systemic, or absorptive,local hormone therapy to achieve immunosuppression. It is still in use within 2 weeks before enrollment.
* Subjects with severe allergic reactions to other monoclonal antibodies.
* The subjects had a central nervous system metastases of clinical symptoms.
* A heart condition or disease that is not well controlled.
* Subjects had active infections.
* Other clinical trials of drugs were used within 4 weeks prior to the first administration.
* The subjects have received other PD-1 antibody therapy or other immunotherapy for PD-1 / PD-L1 or CDK4/6 inhibitor treatment in the past.
* There are other factors lead to patients can not participate in this clinical study by the judgment of the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-01-30 (Estimated); Primary Completion 2020-01-30 (Estimated); Study Completion 2021-01-30 (Estimated)

PRIMARY OUTCOMES:
R0 (resection rate) | 1 week after surgery
  R0 resection rate

SECONDARY OUTCOMES:
ORR | from the first drug administration up to one year
  Objective Response Rate
RFS | from the first drug administration up to one year
  relapse free survival

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Yanqiao, PHD, Principal Investigator — Study Principal Investigator Harbin Medical University Cancer Hosptital